CLINICAL TRIAL: NCT00732901
Title: Project 1: Clinical Neurobiology of Serotonin and Addiction
Brief Title: Clinical Neurobiology of Serotonin and Addiction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HM15289 - 2; P20DA024157 (NIH); DA 024157 (Other)
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2017-06

CONDITIONS: Cocaine Dependence
Keywords: substance abuse; cocaine; impulsivity; serotonin; Remeron; Mirtzapine; Lexapro; Escatilopram
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Impulsive Behavior | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (escitalopram) (Experimental): Escitalopram
  Interventions: Drug: Escitalopram
- B (placebo) (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — Escitalopram: once daily 10 mg on days 1-3, 20 mg on days 4-24 and 10 mg on days 25-28
  Other Names: Lexapro
  Arms: A (escitalopram)
Drug: Placebo — Once daily days 1-28
  Arms: B (placebo)

SUMMARY:
The purpose of this study is to examine the relationship between 5-HT2R function, impulsivity and cue reactivity in cocaine dependent subjects and healthy controls and examine specific effects of escitalopram and mirtazapine on impulsivity and cue reactivity in human cocaine users.

DETAILED DESCRIPTION:
Specific Aim 1: We will test the hypothesis that cocaine-dependent subjects will exhibit greater impulsivity than controls as determined by a battery of impulsivity measures and that impulsivity will be associated with specific profiles of 5-HT2AR and/or 5-HT2CR expression in platelets. We predict that treatment of cocaine-dependent subjects with escitalopram and/or mirtazapine will reduce impulsivity and cocaine-positive urines, in concert with a normalized balance of platelet 5-HT2AR and/or 5-HT2CR expression.

Specific Aim 2: We will test the hypothesis that cocaine-dependent subjects will exhibit greater cue reactivity than controls as determined by a modified Stroop task, and that cue reactivity will be associated with specific profiles of 5-HT2AR and/or 5-HT2CR expression in platelets. We predict that treatment of cocaine-dependent subjects with escitalopram and/or mirtazapine will reduce cue reactivity and cocaine-positive urines, in concert with a normalized balance of platelet 5-HT2AR and/or 5-HT2CR expression.

Specific Aim 3: We will test the hypothesis that specific polymorphisms in the 5-HT2AR and/or 5-HT2CR will predict baseline impulsivity and/or cue reactivity as well as treatment response to serotonergic medications in cocaine-dependent subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non-Drug Abusing Control Subjects: Male and female subjects age 18 to 55 who do not meet current or past DSM-IV criteria for any Axis I disorder including substance abuse or dependence.
* Cocaine Dependent Subjects: Male and female subjects age 18 to 55 who meet current DSM-IV criteria for cocaine dependence.
* Female subjects: a negative pregnancy test.

Exclusion Criteria:

* Non-Drug Abusing Control Subjects:

  1. Current or past DSM-IV Axis I disorder
  2. Any serious non-psychiatric medical illness requiring ongoing medical treatment or which could affect the central nervous system.
  3. Positive HIV test.
  4. For female subjects: a positive pregnancy test or breast feeding.
  5. Concomitant use of prescription medications that could affect the central nervous system.
  6. Active suicidal ideation.
  7. Hamilton Depression or Anxiety Scale score greater than 15
* Cocaine Dependent Subjects:

  1. Current DSM-IV Axis I disorder other than substance abuse/dependence
  2. Current diagnosis of other substance dependence besides cocaine.
  3. Any serious non-psychiatric medical illness requiring ongoing medical treatment or which could affect the central nervous system.
  4. Positive HIV test.
  5. For female subjects: a positive pregnancy test or breast feeding.
  6. Concomitant use of prescription medications that could affect the central nervous system.
  7. Active suicidal ideation.
  8. Subjects within 14 days of discontinuing a monoamine oxidase inhibitor.
  9. Subjects with cardiac arrythmias.
  10. Subjects with known hypersensitivity to escitalopram or citalopram, or mirtazapine
  11. Hamilton Depression or Anxiety Scale score greater than 15.
  12. Current alcohol abuse or dependence.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2008-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- University of Texas Health Science Center-Houston; Substance Abuse Research Clinic, Houston, Texas, United States

REFERENCES:
- [Result] Liu S, Lane SD, Schmitz JM, Waters AJ, Cunningham KA, Moeller FG. Relationship between attentional bias to cocaine-related stimuli and impulsivity in cocaine-dependent subjects. Am J Drug Alcohol Abuse. 2011 Mar;37(2):117-22. doi: 10.3109/00952990.2010.543204. Epub 2011 Jan 5. PMID 21204739
- [Result] Anastasio NC, Liu S, Maili L, Swinford SE, Lane SD, Fox RG, Hamon SC, Nielsen DA, Cunningham KA, Moeller FG. Variation within the serotonin (5-HT) 5-HT(2)C receptor system aligns with vulnerability to cocaine cue reactivity. Transl Psychiatry. 2014 Mar 11;4(3):e369. doi: 10.1038/tp.2013.131. PMID 24618688
- [Result] Liu S, Lane SD, Schmitz JM, Cunningham KA, John VP, Moeller FG. Effects of escitalopram on attentional bias to cocaine-related stimuli and inhibitory control in cocaine-dependent subjects. J Psychopharmacol. 2013 Sep;27(9):801-7. doi: 10.1177/0269881113492898. Epub 2013 Jun 12. PMID 23761390

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment number was the number of participants who signed the informed consent. The Participants who Started in the Participant flow module were number of participants who completed the screening and met inclusion criteria to start medication.
Groups:
- A (Escitalopram): Escitalopram
  Escitalopram: once daily 10 mg on days 1-3, 20 mg on days 4-24 and 10 mg on days 25-28
- B (Placebo): Placebo
  Placebo: once daily for days 1-28
Period: Overall Study
Arm/Group | A (Escitalopram) | B (Placebo)
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A (Escitalopram): Escitalopram: once daily 10 mg on days 1-3, 20 mg on days 4-24 and 10 mg on days 25-28
- B (Placebo): Placebo once daily for days 1-28
- Total: Total of all reporting groups
Arm/Group | A (Escitalopram) | B (Placebo) | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (7.88) | 41.75 (6.65) | 40.01 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 11 | 21
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Immediate Memory Task
Description: The IMT was used to measure impulsivity. The IMT is a continuous performance test. Subjects were instructed to respond on the computer's left mouse button when a five-digit number the target stimulus appeared that was exactly like the preceding stimulus. A catch stimulus was a number that differed only slightly from the preceding number. Only one of the five digits was changed its position and value was determined randomly. Responses errors made to catch stimuli were considered commission errors or 'false alarms'. Immediate Memory Task Commission Errors to catch stimuli were the primary measure of impulsivity in this study. Scale is percentage of overall responses to a catch stimulus that were commission errors, ranging from 0 to 100. Zero would equate to no impulsivity and 100 would equate to 100% impulsive responses.
Time Frame: after acute dose and after chronic administration
Population: Numerical data values are not accessible because PI transferred institutions. See references.
Groups:
- A (Escitalopram): Escitalopram
  Escitalopram: 10 mg daily for days 1-3, 20mg daily for days 4-24, and 10mg daily for days 25-28
- B (Placebo): Placebo
  Placebo: daily for days 1-28
Arm/Group | A (Escitalopram) | B (Placebo)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Attentional Bias as Measured by the Cocaine Stroop Task.
Description: Attentional bias is the difference in reaction time to cocaine related words and neutral words. A slower reaction time indicates greater attentional bias.
Time Frame: 5 weeks of treatment
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | A (Escitalopram) | B (Placebo)
Number analyzed (Participants) | 11 | 12
milliseconds
  Baseline | 90.2 (107.8) | 45.9 (109.2)
  Acute | -8.6 (21.6) | 37.4 (93.8)
  Chronic Day 1 | 56.4 (58.7) | 35.4 (77.9)
  Chronic Day 2 | 45.0 (68.6) | 15.4 (64.5)
  Chronic Day 3 | 23.4 (33.0) | -11.3 (68.0)
  Chronic Day 4 | 63.6 (82.5) | 4.4 (76.2)

3. Secondary Outcome: Cocaine Positive Urines
Description: Number of urine drug screens positive for cocaine metabolite benzoylecgonine.
Time Frame: 5 weeks of treatment
Measure: Number; unit: Positive urine drug screens
Arm/Group | A (Escitalopram) | B (Placebo)
Number analyzed (Participants) | 11 | 12
Positive urine drug screens | 9 | 8

ADVERSE EVENTS:
Arm/Group | A (Escitalopram) | B (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No